CLINICAL TRIAL: NCT03123757
Title: Assessing the Determinants of 6-minute Walk Test and Its Correlation With Quality of Life: A Survey of Older Adults
Brief Title: Assessing the Determinants of 6-minute Walk Test and Its Correlation With Quality of Life
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Precision Health Economics (Other)
Collaborators: Sanofi (Industry)
Responsible Party: Principal Investigator, Jason Shafrin, Principal Investigator, Precision Health Economics
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: Mobility and Quality of Life
Record Dates: First submitted 2017-04-11; First posted 2017-04-21 (Actual); Last update posted 2017-04-21 (Actual); Status verified 2017-04

CONDITIONS: Aged

STUDY DESIGN:
Intervention Model Description: All subjects enrolled in our trial performed the 6-minute walk test and completed an EQ-5D quality of life questionnaire.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention (Other): Patients performed the 6-minute walk test and completed the EQ-5D quality of life questionnaire.
  Interventions: Other: 6 Minute Walk Test; Other: EQ-5D Survey; Other: Short Physical Performance Battery

INTERVENTIONS:
Other: 6 Minute Walk Test — The 6 minute walk test measures the distance walked in 6 minutes without sitting and without the use of a walker or the help of another person (a cane may be used). The walk was conducted in a wide hallway, specifically designed for this type of assessment, with a defined 20-meter course. The subject walked back and forth in the hallway for six minutes and the distance covered was recorded.
Other: EQ-5D Survey — The EQ-5D is a self-reported questionnaire that describes a respondent's health using a descriptive system comprised of five items, each representing a different health dimension (mobility, self-care, usual activities, pain/discomfort, and anxiety/depression). For each dimension, respondents state whether they have no problems, slight problems, moderate problems, severe problems, or are unable to perform the activity.
Other: Short Physical Performance Battery — The SPPB is a brief performance battery based on timed short distance walk, repeated chair stands and balance test administered by trained examiners. The measurement goal for this battery is to assess lower extremity functional limitations, which indicate functional abilities and are a strong measure of risk for future disability.
  Other Names: SPPB

SUMMARY:
This study evaluates the determinants of mobility, measured by the 6-minute walk test, and its correlation with quality of life in near elderly patients.

DETAILED DESCRIPTION:
To evaluate the determinants of mobility an its correlation with quality of life, we conducted a study that evaluated patients ability to perform the 6-minute walk test and their corresponding quality of life measured by the EQ-5D. Cognition was evaluated used the Callahan six-item screener, and additional measures of physical performance were assessed using the Short Physical Performance Battery. Participants disclosed self reported physical function and physical activity. Additionally, other participant characteristics including vital signs, medication history and healthcare utilization were determined as well as social, economic and health related information was collected.

ELIGIBILITY:
Inclusion Criteria:

* Willing to provide informed consent
* Willing to perform the 6-minute walk without the use of a walker, or the assistance of another person.
* Ability to speak and understand English

Exclusion Criteria:

* Medical condition that precludes safe participation in the 6 minute walk test

Ages: 50 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 207 (Actual)
Dates: Start 2015-04-01 (Actual); Primary Completion 2015-08-31 (Actual); Study Completion 2015-08-31 (Actual)

PRIMARY OUTCOMES:
Patient-Reported Quality of Life | On the day of assessment
  Measured using the EQ-5D instrument

SECONDARY OUTCOMES:
Mobility | On the day of assessment
  Measured using the 6-minute walk test

CONTACTS AND LOCATIONS:
Overall Officials: Jason Shafrin, PhD, Principal Investigator — Precision Health Economics

IPD SHARING:
Plan to Share IPD: Undecided